CLINICAL TRIAL: NCT06775756
Title: Phase 3, Prospective, Randomized, Open-Label Study on Simultaneously Reducing Both the Dose and the Irradiated Volume of Cervical Prophylactic Irradiation in Nasopharyngeal Cancer
Brief Title: Reducing Dose and Irradiated Volume in Cervical Prophylactic Irradiation for Nasopharyngeal Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CerviReduce
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental arm receives IMRT to the primary tumor and involved lymph nodes, with a reduced dose and volume of cervical prophylactic irradiation.
  Interventions: Radiation: IMRT with reduced-dose and reduced-volume cervical prophylactic irradiation
- Control Group (No Intervention): The standard arm receives IMRT to the primary tumor and involved lymph nodes, with conventional cervical prophylactic irradiation according to 2024 CSCO guideline. Prescribing dose for CTVn2 was 56Gy/33Fx.

INTERVENTIONS:
Radiation: IMRT with reduced-dose and reduced-volume cervical prophylactic irradiation — For N0 disease, only cover bilateral RPN and level II. For N1 disease, cover ipsilateral involved level plus subsequent level downword, and cover contralateral level RPN and level II. For N2 disease, cover ipsilateral involved level plus subsequent level downword. For N3 disease, cover ipsilateral involved level plus subsequent level downword, and ensuring a 2cm margin below GTVn if GTVn reach or near the sternoclavicular joint. Notably, for unilateral N3, the contralateral neck would only include RPN and level II. Prescribing dose for CTVn2 was 50Gy/33Fx.
  Arms: Experimental Group

SUMMARY:
The purpose of this study is to investigate whether reducing both the dose and the irradiated volume of cervical prophylactic irradiation in patients with nasopharyngeal cancer can maintain efficacy while decreasing toxicity. This will be achieved through a comparison of standard cervical prophylactic irradiation with a reduced-dose and reduced-volume approach.

DETAILED DESCRIPTION:
Patients with non-metastatic nasopharyngeal cancer who are candidates for receiving definitive IMRT are randomly assigned to receive either standard cervical prophylactic irradiation or a reduced-dose and reduced-volume approach. The standard arm receives the conventional dose and volume of irradiation, while the experimental arm receives a lower dose and a smaller irradiated volume. Both groups will undergo intensity-modulated radiotherapy (IMRT) to the primary tumor and involved lymph nodes. The primary endpoint of this study is regional-control (RC), and secondary endpoints include overall survival (OS), local control (LC), distant metastasis-free survival (DMFS), and toxicity. All efficacy analyses will be conducted in the intention-to-treat population, and the safety population will include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic diagnosis (pathologically confirmed by nasopharyngeal biopsy) was nasopharyngeal carcinoma;
2. No distant metastatic;
3. Patients with baseline MRI date of nasopharynx and neck, and completed the first course of treatment in our hospital;
4. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1;
5. Signing informed consent;
6. Follow up regularly and comply with test requirements.

Exclusion Criteria:

1. Disease progression during IMRT;
2. Previous malignancy or other concomitant malignant diseases;
3. The evaluation information of tumor efficacy can not be obtained;
4. Receive blind treatment in other clinical research;
5. Have or are suffering from other malignant tumors within 5 years (except non- melanoma skin cancer or pre-invasive cervical cancer);
6. Serious complications, such as uncontrolled hypertension, coronary heart disease, diabetes, heart failure, etc;
7. Active systemic infection;
8. No or limited capacity for civil conduct;
9. The patient has a physical or mental disorder, and the researcher considers that the patient is unable to fully or fully understand the possible complications of this study;
10. Pregnancy or lactation period;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Regional failure-free survival | 3 years
  The regional relapse-free survival rate will be estimated using Kaplan-Meier method for each arm from the date of randomization to the date of nodal relapse or death from any cause, whichever occurred first. Their differences will be compared between treatment arms using the log-rank test.

SECONDARY OUTCOMES:
Overall Survival | 3 years
  time from the date of the start of chemotherapy to death due to any cause
Local failure-free survival (LFFS) | 3 years
  The duration of time to LFFS was calculated from the date of histological diagnosis until documented treatment local failure or death from any cause.
Distant metastasis-free survival | 3 years
  The distant metastasis-free survival rate will be estimated using Kaplan-Meier
Number of participants with adverse events | 3 years
Incidence of acute and late toxicity | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shaojun Lin, DR, Study Chair — Fujian Cancer Hospital